CLINICAL TRIAL: NCT04069260
Title: A Phase 2, Single Center, Open-Label, Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Daily Subcutaneously Administered ELX-02 in Patients With Nephropathic Cystinosis Bearing One or More CTNS Gene (Cystinosin) Nonsense Mutations
Brief Title: A Phase 2 Study of ELX-02 in Patients With Nephropathic Cystinosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to study design limitations, this study has been discontinued and will not proceed with the 2nd cohort as contemplated in the original protocol.
Sponsor: Eloxx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EL-003
Record Dates: First submitted 2019-08-16; First posted 2019-08-28 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2019-12

CONDITIONS: Genetic Disease; Nonsense Mutation; Cystinosis
Keywords: aminoglycoside; translational read-through; cystinosis; nonsense mutation
MeSH Terms: conditions — Genetic Diseases, Inborn; Cystinosis | interventions — ELX-02

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX-02 (Experimental): Eukaryotic ribosomal selective glycoside (ERSG)
  Interventions: Drug: ELX-02

INTERVENTIONS:
Drug: ELX-02 — ELX-02 is a small molecule, new chemical entity being developed for the treatment of genetic diseases caused by nonsense mutations. ELX-02 is a eukaryotic ribosomal selective glycoside (ERSG).

SUMMARY:
This is a Phase 2 open label study to evaluate the safety, tolerability, PK, and PD of multiple dose levels of SC administered ELX-02 in patients with cystinosis with nonsense mutation in at least one allele.

Six patients will be enrolled in the trial.

The study will comprise of the following periods for each patient:

* A screening period of up to 6 weeks
* A total treatment period of 4 weeks
* A safety follow-up period of 4 weeks after the last treatment

Each patient will receive three escalating doses as follows:

* Treatment period 1: ELX-02 0.5 mg/kg SC daily for 7 days (total dose not to exceed 3.5 mg/kg for this week; the daily dose will be individualized to achieve the target weekly exposure of about 47.5 µg*h/mL)
* Treatment period 2: ELX-02 1.0 mg/kg SC daily for 7 days (total dose not to exceed 7.0 mg/kg for this week; the daily dose will be individualized to achieve the target weekly exposure of about 95 µg*h/mL)
* Treatment period 3: ELX-02 2.0 mg/kg SC daily for 14 days (total dose not to exceed 14 mg/kg for these two weeks; the daily dose will be individualized to achieve the target weekly exposure of about 190 µg*h/mL)

ELIGIBILITY:
Patients must meet all of the following criteria to participate in this study:

1. Male or female patients who, at the time of screening, are 18 years of age or older (Cohort 1) or ≥12 years of age (Cohort 2)
2. A diagnosis of nephropathic cystinosis and biallelic CTNS mutations, including at least one nonsense mutation
3. Patients should have a mild to moderate disease estimated glomerular filtration rate ≥40 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration CKD-EPI formula
4. Body mass index of 19.0 to 30.0 kg/m2. Patients with a lower BMI may be entered into the study at the discretion of the Investigator following consultation with the Sponsor
5. Renal transplant permitted with stable graft function (serum creatinine) for 3 months prior to Screening

Patients with any of the following characteristics/conditions will not be included in the study:

1. Participation in clinical study including administration of any investigational drug or device in the last 30 days or 5 half-lives (whichever is longer) prior to investigational product dosing in the current study
2. Concomitant use of cysteamine bitartrate from 7 days prior to baseline until 7 days following final administration ELX-02
3. An average systolic blood pressure and/or diastolic blood pressure ≥95th percentile for sex, age, and height on 3 or more occasions during the screening period
4. Patients without documented prior aminoglycoside exposure who have a mitochondrial mutation that has been shown to increase sensitivity to aminoglycosides
5. Known relevant allergy or hypersensitivity to aminoglycosides

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
AEs associated with different dose levels of ELX-02 | From the time of first dosing through the follow-up visit, an average of approximately 10 weeks
Area under the plasma concentration curve from time zero to 24 hours (AUC0-24h) | Day 1 of treatment periods 1, 2, and 3
  Full PK profile 12 blood samples over 24 hours
Maximum observed plasma concentration (Cmax) | Day 1 of treatment periods 1, 2, and 3
  Full PK profile 12 blood samples over 24 hours
Observed plasma concentration at 1 hour post dose (C1h) | Days 1, 2, 5, and 7 of treatment periods 1-2; Days 1, 2, 5, 7, 10, and 14 of treatment period 3
  Sparse sampling, blood sampling only, pre-dose and 1 hour post dose
Amount of ELX-02 excreted in urine from 0 to 24 hours (Ae24h) | Day 1 of treatment periods 1, 2, and 3
  6 urine collections over 24 hours
Renal clearance on Day 1 (Ae24h/plasma AUC0-24h) | Day 1 of treatment periods 1, 2, and 3
  6 urine collections over 24 hours

SECONDARY OUTCOMES:
Changes from baseline in WBC cystine levels | Screening; Days 1, 2, 5, and 7 of treatment periods 1-2; Days 1, 2, 5, 7, 10, and 14 of treatment period 3, and 4-week safety follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goodyer, MD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- See also: Eloxx Pharmaceuticals Website — http://www.eloxxpharma.com